CLINICAL TRIAL: NCT04022304
Title: A Randomised, Double-blind, Three-period, Partially Replicated Crossover, Euglycaemic Glucose Clamp Study in Healthy Volunteers to Demonstrate Pharmacokinetic and Pharmacodynamic Similarity of Biocon Insulin N and Humulin® N
Brief Title: Comparision of Pharmacokinetic and Pharmacodynamic of Biocon Insulin N and Humulin® N
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biocon Limited (Industry)
Collaborators: Profil Institut für Stoffwechselforschung GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: EQN
Record Dates: First submitted 2019-06-29; First posted 2019-07-17 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Healthy Volunteer
Keywords: Recombinant Human Insulin N (rhi N)

STUDY DESIGN:
Intervention Model Description: Partially replicated design, crossover trial
Who Masked: Participant, Investigator
Masking Description: Double blind study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Sequence: Humulin® N- Biocon Insulin N-Humulin® N (Experimental): Period 1: 0.4 IU/kg of Humulin® N (100 IU/mL) administered once subcutaneously.
  Period 2: 0.4 IU/kg of Biocon Insulin N (100 IU/mL) administered once subcutaneously.
  Period 3: 0.4 IU/kg of Humulin® N (100 IU/mL) administered once subcutaneously.
  The treatment periods will be separated by 5-7 days
  Interventions: Biological: Biocon Insulin N; Biological: Humulin® N
- Sequence: Biocon Insulin N- Humulin® N- Humulin® N (Experimental): Period 1: 0.4 IU/kg of Biocon Insulin N (100 IU/mL) administered once subcutaneously.
  Period 2: 0.4 IU/kg of Humulin® N(100 IU/mL) administered once subcutaneously.
  Period 3: 0.4 IU/kg of Humulin® N (100 IU/mL) administered once subcutaneously.
  The treatment periods will be separated by 5-7 days
  Interventions: Biological: Biocon Insulin N; Biological: Humulin® N
- Sequence: Humulin® N- Humulin® N-Biocon Insulin N (Experimental): Period 1: 0.4 IU/kg of Humulin® N(100 IU/mL) administered once subcutaneously.
  Period 2: 0.4 IU/kg of Humulin® N (100 IU/mL) administered once subcutaneously.
  Period 3: 0.4 IU/kg of Biocon Insulin N (100 IU/mL) administered once subcutaneously.
  The treatment periods will be separated by 5-7 days
  Interventions: Biological: Biocon Insulin N; Biological: Humulin® N
- Sequence: Biocon Insulin N- Humulin® N- Biocon Insulin N (Experimental): Period 1: 0.4 IU/kg of Biocon Insulin N (100 IU/mL) administered once subcutaneously.
  Period 2: 0.4 IU/kg of Humulin® N (100 IU/mL) administered once subcutaneously.
  Period 3: 0.4 IU/kg of Biocon Insulin N (100 IU/mL) administered once subcutaneously.
  The treatment periods will be separated by 5-7 days
  Interventions: Biological: Biocon Insulin N; Biological: Humulin® N
- Sequence: Humulin® N-Biocon Insulin N- Biocon Insulin N (Experimental): Period 1: 0.4 IU/kg of Humulin® N (100 IU/mL) administered once subcutaneously.
  Period 2: 0.4 IU/kg of Biocon Insulin N (100 IU/mL) administered once subcutaneously.
  Period 3: 0.4 IU/kg of Biocon Insulin N (100 IU/mL) administered once subcutaneously.
  The treatment periods will be separated by 5-7 days
  Interventions: Biological: Biocon Insulin N; Biological: Humulin® N
- Sequence: Biocon Insulin N- Biocon Insulin N-Humulin® N (Experimental): Period 1: 0.4 IU/kg of Biocon Insulin N (100 IU/mL) administered once subcutaneously.
  Period 2: 0.4 IU/kg of Biocon Insulin N (100 IU/mL) administered once subcutaneously.
  Period 3: 0.4 IU/kg of Humulin® N (100 IU/mL) administered once subcutaneously.
  The treatment periods will be separated by 5-7 days
  Interventions: Biological: Biocon Insulin N; Biological: Humulin® N

INTERVENTIONS:
Biological: Biocon Insulin N — Biocon Insulin N is an intermediate-acting isophane suspension of human insulin produced by recombinant deoxyribonucleic acid(rDNA) technology utilizing Pichia pastoris (yeast).
Biological: Humulin® N — Humulin® N (human insulin [recombinant deoxyribonucleic acid origin] isophane suspension) is an intermediate-acting human isophane insulin. Humulin® N is a suspension of crystals produced from combining human insulin and protamine sulphate.

SUMMARY:
Single-centre, randomised, double-blind, three-period, six-sequence, partially replicated design, crossover trial in healthy subjects

DETAILED DESCRIPTION:
The present study is designed to demonstrate pharmacokinetic and pharmacodynamic equivalence of Biocon Insulin N with Humulin® N in healthy subjects.

The treatment consists of one single dose of the test or reference product, administered during each of the three study periods, separated by 5-7 days between each dosing. The planned trial duration for each subject is about 17 to 43 days. Eligible subjects will undergo three euglycaemic clamp examinations (each of 24 hours duration).

Depending on the sequence in which a particular subject is randomized, each subject will either undergo two clamps with administration of test product plus one clamp with administration of reference product, or, two clamps with administration of reference product plus one clamp with administration of test product, in random order.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and post-menopausal female subjects. Post-menopausal defined as 12 months of no menses without an alternative medical cause and confirmed by a follicle stimulating hormone (FSH) level in the post-menopausal range (>= 25.8 IU/L).
2. Age between 18 and 55 years, both inclusive
3. Body mass index between 18.5 and 29.0 kg/m^2, both inclusive.
4. Fasting plasma glucose concentration <= 100 mg/dl.
5. Considered generally healthy upon completion of medical history and screening safety assessments, as judged by the Investigator.

Exclusion Criteria:

1. Known or suspected hypersensitivity to Investigational Medicinal products (IMP(s)) or related products.
2. Systolic blood pressure < 95 mmHg or >140 mmHg and/or diastolic blood pressure < 50 mm Hg or >90 mmHg after resting for at least 5 minutes in supine position (excluding white-coat hypertension; therefore, a repeat test showing results within range will be acceptable).
3. Pulse rate at rest outside the range of 50-90 beats per minute.
4. Receipt of any medicinal product in clinical development within 30 days or five times its half-life (whichever is longer) before randomisation.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2019-06-15 (Actual); Primary Completion 2019-12-21 (Actual); Study Completion 2019-12-27 (Actual)

PRIMARY OUTCOMES:
Primary PK endpoint: area under the insulin concentration curve(AUCins).0-24h | 0-24hour
  area under the insulin concentration curve
Primary PK endpoint: maximum observed insulin concentration(Cins.max) | 0-24hour
  maximum observed insulin concentration
PD endpoint:area under the glucose infusion rate curve(AUCGIR)0-24h | 0-24hour
  area under the glucose infusion rate curve
PD endpoint:maximum observed glucose infusion rate (GIRmax) | 0-24hour
  maximum observed glucose infusion rate

SECONDARY OUTCOMES:
Secondary PK endpoint: area under the insulin concentration-time curve(AUCins).0-infinity | 0-24 hours
  area under the insulin concentration-time curve
Secondary PK endpoint: area under the insulin concentration-time curve(AUCins).0-12h | 0-12hour
  area under the insulin concentration-time curve
Secondary PK endpoint: area under the insulin concentration-time curve(AUCins).12-24h | 12-24hour
  area under the insulin concentration-time curve
Secondary PK endpoint:time to maximum observed insulin concentration (tmax.ins) | 0-24 hours
  time to maximum observed insulin concentration
Secondary PK endpoint:terminal elimination rate constant of insulin (λz) | 0-24 hours
  terminal elimination rate constant of insulin
Secondary PK endpoint: terminal elimination half-life (t½) | 0-24 hours
  terminal elimination half-life calculated as t½=ln2/λz
Secondary PK endpoint: time(t)50%-INS(early) | 0-24 hours
  time to half-maximum before Cmax
Secondary PK endpoint: time(t)50%-INS(late) | 0-24 hours
  time to half-maximum after Cmax
Secondary PD endpoint: areas under the glucose infusion rate curve(AUCGIR).0-12h | 0-12hours
  areas under the glucose infusion rate curve
Secondary PD endpoint: areas under the glucose infusion rate curve(AUCGIR).12-24h | 12-24hours
  areas under the glucose infusion rate curve
Secondary PD endpoint: time to maximum glucose infusion rate(tmax.GIR) | 0-24 hours
  time to maximum glucose infusion rate
Secondary PD endpoint:time to half-maximum glucose infusion rate before GIRmax (tGIR.50%-early) | 0-24 hours
  time to half-maximum glucose infusion rate before GIRmax
Secondary PD endpoint: time to half-maximum glucose infusion rate after GIRmax (tGIR.50%-late) | 0-24 hours
  time to half-maximum glucose infusion rate after GIRmax
Secondary PD endpoint: Onset of action | 0-24 hours
  time from trial product administration until blood glucose concentration has decreased at least 5 mg/dL from baseline, where baseline is defined as the mean of blood glucose levels from -6, -4, and -2 minutes before trial product administration as measured by ClampArt(name of Clamp Devise))

OTHER OUTCOMES:
Safety endpoint: Number of subjects with Adverse Events (AEs), clinically significant changes in Physical examination, Vital signs. Local tolerability/ Injection site reactions | First dose to followup period (Total duration: 21 days approximate)
  Number of subjects with Adverse Events (AEs), clinically significant changes in Physical examination, Vital signs.
  Local tolerability/ Injection site reactions
Safety endpoint: Number of subjects with clinically significant changes in Laboratory safety parameters, Electrocardiogram (ECG) | Screening and Follow-up period (Total duration: 42 days approximate)
  Number of subjects with clinically significant changes in Laboratory safety parameters.
  Number of subjects with clinically significant changes in Electrocardiogram (ECG)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Grit Andersen, Principal Investigator — Profil Institut für Stoffwechselforschung GmbH Hellersbergstraße 9]
Locations (1):
- Profil Institut für Stoffwechselforschung GmbH, Neuss, Germany